CLINICAL TRIAL: NCT03997500
Title: Prophylactic Norepinephrine Infusion for Spinal Hypotension and Inferior Vena Cava Collapsibility Index During Cesarean Delivery: a Randomized Double Blinded Controlled Study
Brief Title: Prophylactic Norepinephrine Infusion for Spinal Hypotension and Inferior Vena Cava Collapsibility Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Yi Chen
Record Dates: First submitted 2019-05-28; First posted 2019-06-25 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-05

CONDITIONS: Adverse Effect
Keywords: Norepinephrine; Hypotension; Inferior Vena Cava Collapsibility Index; Cesarean Delivery
MeSH Terms: conditions — Hypotension | interventions — Saline Solution; Norepinephrine; Vasoconstrictor Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal saline (Placebo Comparator): Simultaneous with subarachnoid block, a bolus of normal saline was given followed by normal saline infusion
  Interventions: Drug: normal saline
- Norepinephrine (Experimental): Simultaneous with subarachnoid block, a bolus of norepinephrine was given followed by norepinephrine infusion
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: normal saline — a bolus of normal saline was given followed by normal saline infusion
  Other Names: NS
  Arms: Normal saline
Drug: Norepinephrine — a bolus of norepinephrine was given followed by norepinephrine infusion
  Other Names: Vasopressors
  Arms: Norepinephrine

SUMMARY:
The purpose of this study is to investigate the preventive effect of norepinephrine on post-spinal hypotension and the effect of norepinephrine on inferior vena cava collapsibility index (IVC-CI).

DETAILED DESCRIPTION:
Post-spinal hypotension is a frequent complication during spinal anesthesia for cesarean delivery. It affects nearly 50-60% of patients without appropriately treat. Vasopressors has been highly recommended for routine prevention and/or treatment of post-spinal hypotension. Norepinephrine is new vasopressor that has been suggested as a potential alternative to phenylephrine and was recently introduced in obstetric anesthesia because of the minimal cardiac depressant effect. The purpose of this study is to investigate the preventive effect of norepinephrine on post-spinal hypotension and the effect on inferior vena cava collapsibility index (IVC-CI).

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for elective cesarean delivery under spinal anesthesia
* Full-term, singleton, pregnant women

Exclusion Criteria:

* Height of no more than 150 centimeters
* Body weight greater than 100 kg or BMI greater than 30
* Labor analgesia had been performed
* Contraindication of spinal or epidural anesthesia
* Eclampsia or chronic hypertension or baseline blood pressure ≥160mmHg
* Hemoglobin <7g/dl
* Fetal distress or known abnormal fetal development
* Severe vascular disease
* Diabetes mellitus or cardiovascular disease or nervous system disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of hypotension | 1 to 20 minutes after subarachnoid block
  SBP decreased to <80% of the baseline value
Inferior vena cava collapsibility index | 5 to 20 minutes after subarachnoid block
  CI = (dIVCmax - dIVCmin)/dIVCmax

SECONDARY OUTCOMES:
The incidence of nausea and vomiting | 1 to 20 minutes after subarachnoid block
  Presence of nausea and vomiting in patients after subarachnoid block
The incidence of bradycardia | 1 to 20 minutes after subarachnoid block
  Heart rate less than 55 bpm
Incidence of hypertension | 1 to 20 minutes after subarachnoid block
  Systolic blood pressure at or above 120% of baseline
Arterial base excess of fetal vein blood | Immediately after delivery
  From umbilical vein blood gases
Pressure of oxygen of fetal vein blood | Immediately after delivery
  From umbilical vein blood gases
pH value of fetal vein blood | Immediately after delivery
  From umbilical vein blood gases
Number of rescue norepinephrine | Immediately to 20 minutes after subarachnoid block
  a bolus of norepinephrine was given when SBP decreased to <80% of the baseline value
APGAR score | 1min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 10min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, Dr., Study Chair — xinlini6@yahoo.com
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No